CLINICAL TRIAL: NCT03518840
Title: The Predictive Value of the Active Straight Leg Raise on the Efficacy of a Sacroiliac Joint Belt in Posterior Pelvic Girdle Pain During Pregnancy
Brief Title: Predictive Value of the Active Straight Leg Raise on the Efficacy of a SJB in Posterior PGP During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Colleen M. Fitzgerald, MD, MS, M.D. Associate Professor, Loyola University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 210146
Record Dates: First submitted 2018-04-10; First posted 2018-05-08 (Actual); Results first posted 2020-10-28 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Intervention Model Description: All patients receive an SIJ belt.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sacroiliac Joint Belt (Other): All patients will receive and be fitted by the PI with an SIJ belt.
  Interventions: Device: SIJ Belt

INTERVENTIONS:
Device: SIJ Belt — Support Belts

SUMMARY:
During pregnancy, women often experience musculoskeletal pain, specifically in their low back and/or pelvic girdle. Pelvic girdle pain (PGP) is defined as pain between the posterior iliac crest and gluteal fold, particularly in the region of the sacroiliac joint (SIJ)1. Although it is often referred to as "sciatica". PGP in pregnancy is common with prevalence estimates of 45%2. Previous studies have found that one third of patients will rate their PGP intensity as severe, leading to functional impairments. Functional disabilities include sitting, walking, and standing; thus, significantly impacting the ability of patients to perform routine daily activities. This pain has been reported to develop as early as 17-19 weeks' gestation, lasting up to 3 months postpartum; with a peak incidence of 24-36 weeks.

The etiology of PGP in pregnant women is still not fully understood, largely due to the complex interactions between bone, ligaments, fascia, and muscles in the pelvic joints3. Some studies suggest the increased mobility of the joints in the pelvic girdle during pregnancy due to relaxing cause a lack of stabilization in the sacroiliac region, which results in pain4. Thus, it is hypothesized that providing stabilization of the joints with an external force, such as a maternity or SIJ belt, will improve pain.

DETAILED DESCRIPTION:
During pregnancy, women often experience musculoskeletal pain, specifically in their low back and/or pelvic girdle. Pelvic girdle pain (PGP) is defined as pain between the posterior iliac crest and gluteal fold, particularly in the region of the sacroiliac joint (SIJ)1. Although it is often referred to as "sciatica". PGP in pregnancy is common with prevalence estimates of 45%2. Previous studies have found that one third of patients will rate their PGP intensity as severe, leading to functional impairments. Functional disabilities include sitting, walking, and standing; thus, significantly impacting the ability of patients to perform routine daily activities. This pain has been reported to develop as early as 17-19 weeks' gestation, lasting up to 3 months postpartum; with a peak incidence of 24-36 weeks.

The etiology of PGP in pregnant women is still not fully understood, largely due to the complex interactions between bone, ligaments, fascia, and muscles in the pelvic joints3. Some studies suggest the increased mobility of the joints in the pelvic girdle during pregnancy due to relaxing cause a lack of stabilization in the sacroiliac region, which results in pain4. Thus, it is hypothesized that providing stabilization of the joints with an external force, such as a maternity or SIJ belt, will improve pain.

Clinically, pelvic belts are often used as a part of a multimodal approach to reduce PGP alongside other conservative treatments such as analgesics and physical therapy, or more alternative treatments such as acupuncture5. This makes it difficult to determine their individual effect on pain reduction. Further confounding this issue are variations in physician counseling, physical therapy regimens, and analgesic usage. Moreover, several support belts have been designed that vary in padding size, flexibility, and site of application5-7. Among these belts, it has not yet been identified which belt is most beneficial regarding pain reduction and patient tolerance5. Previous studies have found benefit in short term use (3-6 weeks) of maternity belts, providing women with improved pain and function compared to exercise or no intervention7. Pelvic belts are a cost-effective option to treating PGP, and more specifically SIJ pain, yet studies are limited regarding the effect they have on SIJ mobility and pain reduction8 and more specifically determining what clinically predicts those who will benefit most from an SIJ belt.

The active straight leg raise test originally described by Mens is an examination maneuver that measures functional mobility and has been correlated with pregnancy related PGP (cite). Anecdotally, our clinical team has observed that women who benefit from compression during the second part of the test, seem to benefit most from the use of an SIJ belt. Having a simple test for obstetric providers to perform in pregnant women with pain would be informative in determining who might benefit most from an SIJ belt. Hence our study seeks to investigate the following aims:

ELIGIBILITY:
Inclusion Criteria:

* English speaking pregnant women presenting in their second or third trimester with posterior PGP. Trimester will be determined from date of last menses or ultrasound date.
* Pain must be between the upper level of the iliac crests and the gluteal folds in conjunction with or separately from pain in the pubic symphysis and influenced by position and locomotion
* ASLR score between 2-10

Exclusion Criteria:

* Non-English speaking pregnant women <18 or >50 years old
* Women presenting with PGP in the first trimester (<13 weeks gestation)
* Women with pubic symphysis (anterior) pain alone
* Pain above the upper level of the iliac crest
* ASLR total score of <2
* History of lumbar or pelvic fracture, neoplasm, inflammatory disease, active urogenital infection or active gastrointestinal illness, previous surgery of the lumbar spine, pelvic girdle, hip joint or femur
* History or signs of radiculopathy or other systemic neurologic disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Fitzgerald, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Health System, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Wu WH, Meijer OG, Uegaki K, Mens JM, van Dieen JH, Wuisman PI, Ostgaard HC. Pregnancy-related pelvic girdle pain (PPP), I: Terminology, clinical presentation, and prevalence. Eur Spine J. 2004 Nov;13(7):575-89. doi: 10.1007/s00586-003-0615-y. Epub 2004 Aug 27. PMID 15338362
- [Background] Ekman EF, Koman LA. Acute pain following musculoskeletal injuries and orthopaedic surgery: mechanisms and management. Instr Course Lect. 2005;54:21-33. PMID 15948432
- [Background] Kristiansson P, Svardsudd K, von Schoultz B. Serum relaxin, symphyseal pain, and back pain during pregnancy. Am J Obstet Gynecol. 1996 Nov;175(5):1342-7. doi: 10.1016/s0002-9378(96)70052-2. PMID 8942512
- [Background] Flack NA, Hay-Smith EJ, Stringer MD, Gray AR, Woodley SJ. Adherence, tolerance and effectiveness of two different pelvic support belts as a treatment for pregnancy-related symphyseal pain - a pilot randomized trial. BMC Pregnancy Childbirth. 2015 Feb 15;15:36. doi: 10.1186/s12884-015-0468-5. PMID 25885585
- [Background] Kordi R, Abolhasani M, Rostami M, Hantoushzadeh S, Mansournia MA, Vasheghani-Farahani F. Comparison between the effect of lumbopelvic belt and home based pelvic stabilizing exercise on pregnant women with pelvic girdle pain; a randomized controlled trial. J Back Musculoskelet Rehabil. 2013;26(2):133-9. doi: 10.3233/BMR-2012-00357. PMID 23640314
- [Background] Mens JM. Does a pelvic belt reduce hip adduction weakness in pregnancy-related posterior pelvic girdle pain? A case-control study. Eur J Phys Rehabil Med. 2017 Aug;53(4):575-581. doi: 10.23736/S1973-9087.17.04442-2. Epub 2017 Mar 1. PMID 28251846
- [Background] Soisson O, Lube J, Germano A, Hammer KH, Josten C, Sichting F, Winkler D, Milani TL, Hammer N. Pelvic belt effects on pelvic morphometry, muscle activity and body balance in patients with sacroiliac joint dysfunction. PLoS One. 2015 Mar 17;10(3):e0116739. doi: 10.1371/journal.pone.0116739. eCollection 2015. PMID 25781325
- [Derived] Fitzgerald CM, Bennis S, Marcotte ML, Shannon MB, Iqbal S, Adams WH. The impact of a sacroiliac joint belt on function and pain using the active straight leg raise in pregnancy-related pelvic girdle pain. PM R. 2022 Jan;14(1):19-29. doi: 10.1002/pmrj.12591. Epub 2021 May 20. PMID 33745213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from November 2017 through June 2019 (20 months) from a tertiary care female pelvic medicine and reconstructive surgery practice.
Groups:
- Sacroiliac Joint Belt: All patients receive an SIJ belt
Period: Overall Study
Arm/Group | Sacroiliac Joint Belt
Started | 63
Completed | 57
Not Completed | 6
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Sacroiliac Joint Belt
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.94 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 13
  Race: White | 27
  Race: Other | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63
Employment [Count of Participants; unit: Participants]
  Employed | 42
  Stay at home parent | 16
  Unemployed | 5
Previous mode of delivery [Count of Participants; unit: Participants]
  Vaginal | 34
  C-section | 10
  Both | 2
  Not reported | 17
Previous abdominal surgery [Count of Participants; unit: Participants]
  No | 49
  Yes | 13
  Not reported | 1
History of low back pain [Count of Participants; unit: Participants]
  No | 41
  Yes | 22
Prior physical therapy for lower back pain [Count of Participants; unit: Participants]
  No | 59
  Yes | 4
Prior pelvic pain [Count of Participants; unit: Participants]
  No | 52
  Yes | 11
Physical activity level [Count of Participants; unit: Participants]
  Not physically active | 10
  Mildly physically active | 29
  Moderately physically active | 22
  Extremely physically active | 2
Smoker status [Count of Participants; unit: Participants]
  Non-smoker | 43
  Smoker | 20
History of depression [Count of Participants; unit: Participants]
  No | 52
  Yes | 11
History of anxiety [Count of Participants; unit: Participants]
  No | 52
  Yes | 11

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Functioning on the Active Straight Leg Rise (ASLR) Scale at 4 Weeks.
Description: The ASLR scale is an assessment of the functioning level of a patient's affected leg. It ranges from 0 to 5 with higher values indicating greater impairment.
Time Frame: Baseline and 4 weeks
Population: Sixty-three women who signed an informed consent document were available at baseline and 52 women returning for the week 4 follow-up visit completed the ASLR assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: All patients received an SIJ belt and had their ASLR score recorded at baseline
- Week 4: At week 4, 52 women returning completed the ASLR assessment
Arm/Group | Baseline | Week 4
Number analyzed (Participants) | 63 | 52
score on a scale | 4.87 (1.85) | 2.92 (2.43)
Statistical Analysis 1: Comparison: Baseline vs Week 4; The null hypothesis is that there is no change in the baseline ASLR score following four weeks of SIJ belt therapy; Test type: Superiority; p < .001, paired t-test, 2 sided; Mean Difference (Final Values) = -1.9615, 95% CI 2-sided [-2.6299 to -1.2932], Standard Error of Mean 0.3329

2. Secondary Outcome: Change From Baseline in Pain on the Numeric Rating Scale (NRS) at 4 Weeks
Description: The NRS is a pain assessment scale ranging from 0 to 10, where 0 represents "No Pain", 5 represents "Moderate Pain", and a value of 10 represents the "Worst Possible Pain".
Time Frame: Baseline and 4 weeks
Population: Sixty-three women who signed an informed consent document were available at baseline and 57 women returning for the week 4 follow-up visit completed the NRS.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: All patients received an SIJ belt and had their pain score recorded at baseline
- Week 4: At week 4, 57 women completed the NRS assessment
Arm/Group | Baseline | Week 4
Number analyzed (Participants) | 63 | 57
score on a scale | 6.10 (1.93) | 4.18 (2.28)
Statistical Analysis 1: Comparison: Baseline vs Week 4; The null hypothesis is that there is no change in the baseline NRS score following four weeks of SIJ belt therapy; Test type: Superiority; p < .001, paired t-test, 2 sided; Median Difference (Final Values) = -1.9474, 95% CI 2-sided [-2.6190 to -1.2757], Standard Error of Mean 0.3353

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for six weeks
Arm/Group | Sacroiliac Joint Belt
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sacroiliac Joint Belt (N=63)
Pinched nerve (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT03518840/Prot_SAP_001.pdf
  • Informed Consent Form (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT03518840/ICF_002.pdf